CLINICAL TRIAL: NCT00336557
Title: A Randomized, Controlled, Open-Label Parallel Group Study to Evaluate the Effect of Regularly Scheduled Neutralizing Antibody Testing on Treatment Patterns Versus Usual Care in High-Dose Interferon Treated Patients
Brief Title: Determine Impact of Multiple NAb Tests on Treatment Compared to Usual Care of MS Patients on High-dose IFN Therapy
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PM028
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Sclerosis
Keywords: High-Dose Interferon; Neutralizing Antibodies
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood drawn for a Binding Antibody (BAb) and Neutralizing Antibody (NAb) test.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Regularly Scheduled NAb Testing Arm: Subjects will be scheduled for 5 study visits over the course of 12 months and any NAbs test results will be available to the investigator during the study.
  Interventions: Procedure: NAbs testing
- Usual Care Arm: Subjects will be scheduled for 2 study visits over the course of 12 months and any NAbs test results will be unknown by the investigator until the conclusion of the subject's study participation.

INTERVENTIONS:
Procedure: NAbs testing — blood drawn for a Binding Antibody (BAb) and Neutralizing Antibody (NAb) test.
  Groups: Regularly Scheduled NAb Testing Arm

SUMMARY:
An observational study to determine the impact of multiple neutralizing antibody (NAb) tests on treatment patterns compared to the usual care of MS patients receiving high-dose IFN therapy.

DETAILED DESCRIPTION:
An observational study to determine the impact of multiple neutralizing antibody (NAb) tests on treatment patterns compared to the usual care of MS patients receiving high-dose IFN therapy.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent.
* Male or female, 18 years of age or older, with a diagnosis of MS.

Exclusion Criteria:

* Has been on oral or parenteral corticosteroid therapy within the two weeks prior to the Baseline Visit.
* Has been treated with immunoglobulins (IgG) or plasmapheresis within the last six months.
* Has any condition which the investigator or nurse feels may interfere with participation in the study or with assessments for the full duration of the study.
* Previously participated in this study.
* Has received an experimental drug in the last thirty (30) days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have been on high-dose Interferon (IFN) for 1 to 4 years
Sampling Method: Probability Sample
Enrollment: 1230 (Actual)
Dates: Start 2006-07; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects whose high dose IFN therapy had changed in the regularly scheduled NAbs testing arm versus the Usual Care Arm | 1 year

SECONDARY OUTCOMES:
The nature of any therapy/management change in each arm | 1 year
Reason for change in therapy/management | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Glenski, PharmD, Study Chair — Teva Neuroscience, Inc.
Locations (49):
- United States (49):
  - Phoenix Neurological Associates, LTD, Phoenix, Arizona
  - East Bay Physicians Medical Group, Berkley, California
  - Neuro-Pain Medical Center, Fresno, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - University of Southern California, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - Neurology Clinic of Marin, San Anselmo, California
  - Colorado Springs Neurological Associates, PC, Colorado Springs, Colorado
  - Colorado Neurosurgery, Engelwood, Colorado
  - The Emery Neuroscience Center, Fort Lauderdale, Florida
  - Neurology Associates, PA, Maitland, Florida
  - Collier Neurologic Specialitsts, Naples, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Medical College of Georgia Augusta MS Center, Augusta, Georgia
  - Carle Clinic Association, Urbana, Illinois
  - Neurology Associates, Hopedale, Massachusetts
  - Lahey Clinic, Lexinton, Massachusetts
  - South Shores Neurology Associates, INC, South Weymouth, Massachusetts
  - Michigan Neurology Associates, Saint Clair Shores, Michigan
  - Mankato Clinic, Mankato, Minnesota
  - Columbia Center for Neurology and MS, Columbia, Missouri
  - St John's Mercy Medical Center, St Louis, Missouri
  - Advanced Neurology Specialist, Great Falls, Montana
  - Creighton University Department of Neurology, Bellvue, Nebraska
  - The Neuroscience Center of Northern NJ, Morristown, New Jersey
  - Neurology Associates of Albany, P.C., Albany, New York
  - NYU Hospital for Join Diseases, MS Center, New York, New York
  - Comprehensive MS Care Clinic at South Shore Neurology, Patchogue, New York
  - Rochester Multiple Sclerosis Center, Rochester, New York
  - Asheville Neurology Specialist, PA, Asheville, North Carolina
  - East Carolina Neurology, Greenville, North Carolina
  - Alliance for Neuro Research, LLC Absher Neurology, Greenville, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Central Carolina Neurology & Sleep, Salisbury, North Carolina
  - NeuroCare Center, Canton, Ohio
  - Neurology Specialists, Inc, Dayton, Ohio
  - Oak Clinic, Uniontown, Ohio
  - Medford Neurological Clinic,Inc, Medford, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Neurology Associates of Monroe County, East Stroudsburg, Pennsylvania
  - North Shore Clinical Associates, Erie, Pennsylvania
  - NeuroHealth, INC, Warwick, Rhode Island
  - Mid-South Physicians, Germantown, Tennessee
  - Central Texas Neurology, Round Rock, Texas
  - Neurology Center of San Antonio, P.A., San Antonio, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - Rocky Mountain Multiple Sclerosis Clinic, Salt Lake City, Utah
  - Dean Health System, Madison, Wisconsin